CLINICAL TRIAL: NCT03559075
Title: Assessing Caregiver's Confidence in the Use of Topical Corticosteroids for a Child's Atopic Dermatitis
Brief Title: Clinical vs. Anecdotal Evidence - Pediatric Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00051332
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2018-09

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema; children
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Group 1: Participants will be randomized into group 1 to be queried about their comfort with medication for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.
- Group 2: Participants will be randomized into group 2 to be queried about their comfort with medication for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.
- Group 3: Participants will be randomized into group 3 to be queried about their comfort with medication for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.
- Group 4: Participants will be randomized into group 4 to be queried about their comfort with a topical steroid for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.
- Group 5: Participants will be randomized into group 5 to be queried about their comfort with a topical steroid for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.
- Group 6: Participants will be randomized into group 6 to be queried about their comfort with a topical steroid for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.
- Group 7: Participants will be randomized into group 7 to be queried about their comfort with medication for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.
- Group 8: Participants will be randomized into group 8 to be queried about their comfort with medication for treating their child's atopic dermatitis after hearing varying amounts of information about the treatment.

SUMMARY:
In dermatology, topical anti-inflammatory medications, such as corticosteroids, are the mainstay treatment of managing patients with atopic dermatitis. However, caregivers are often apprehensive about choosing a topical steroid for a variety of reasons. Many caregivers are not aware that clinical trial evidence for these medications exist, and instead may rely on anecdotal evidence in choosing to take these medications. Because fear of the drug is inherently subjective, it can be modified with appropriate reassurance and presentation of evidence. The goal of the study is to learn whether caregivers are more confident in treating a child's atopic dermatitis after being presented with varying amounts of information.

DETAILED DESCRIPTION:
Atopic dermatitis is the most common chronic, inflammatory dermatologic condition in young children, with a prevalence approaching 25% in some countries. Topical corticosteroids, the mainstay treatment in managing atopic dermatitis, generally function to decrease inflammation and suppress the immune response. Topical corticosteroids are grouped into distinct categories based on their degree of potency, including very high potency (Clobetasol propionate), high potency (triamcinolone acetonide), medium potency (fluocinonide), and low potency agents (desonide).

Caregivers are often apprehensive about choosing a topical steroid for a variety of reasons. These include hearing negative information about the drug from friends or family, being nervous about treatment, or seeing the drug or its side effects negatively portrayed in the media. Many parents/caregivers are not aware that clinical trial evidence for these medications exist, and instead may rely on anecdotal evidence in choosing to take these medications.

Because fear of the drug is inherently subjective, it can be modified with appropriate reassurance and presentation of evidence. By understanding what kind of information will allow caregivers to be confident in their decision to use a topical corticosteroid, dermatologists may improve treatment adherence and outcomes. The goal of the study is to learn whether caregivers are more confident in treating a child's atopic dermatitis after being presented with varying amounts of information about the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Caregiver of an individual age <1-17 years old
* Subjects with a working knowledge of English

Exclusion Criteria:

* Parent/Caregiver of an individual 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects meeting the following characteristics will be eligible to participate: caregiver of an individual age <1-17, and possessing a working knowledge of English.
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Survey responses on "willingness to treat" | 1 day
  Groups 1, 2, and 3 will be compared to assess whether caregivers are more willing to use a medication to manage their child's atopic dermatitis if presented with clinical trial evidence, anecdotal evidence, or both. Groups 4, 5, and 6 will be compared to assess whether caregivers are more willing to use a topical steroid to manage their child's atopic dermatitis if presented with clinical trial evidence, anecdotal evidence, or both. The results from groups 1, 2, and 3 will then be compared to the results from groups 4, 5, and 6 to assess whether the use of the word "steroid" impacts the caregiver's willingness to treat.
Survey responses on "willingness to treat with doctor's recommended medication" | 1 day
  Groups 7 and 8 will be compared to assess how caregiver's willingness to treat with a doctor's recommended medication is impacted by the exclusion of anecdotal evidence, clinical trial evidence, or both.

CONTACTS AND LOCATIONS:
Overall Officials: Stevan Feldman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buhrmester M, Kwang T, Gosling SD. Amazon's Mechanical Turk: A New Source of Inexpensive, Yet High-Quality, Data? Perspect Psychol Sci. 2011 Jan;6(1):3-5. doi: 10.1177/1745691610393980. Epub 2011 Feb 3. PMID 26162106